CLINICAL TRIAL: NCT07286552
Title: Noninvasive Breathing Pattern Monitoring in Patients With Acute Respiratory Failure Secondary to Pneumonia Requiring Hospital Admission: Differences Based on Clinical Outcomes
Brief Title: Breathing Pattern Description in Pneumonia Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Consorci Sanitari Integral (Other)
Responsible Party: Sponsor
Other Study IDs: MAR202122-30
Record Dates: First submitted 2025-08-11; First posted 2025-12-16 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: Acute Respiratory Failure (ARF)
Keywords: Respiratory failure; coronavirus infection; bacterial pneumonia
MeSH Terms: conditions — Respiratory Insufficiency; Coronavirus Infections; Pneumonia, Bacterial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with pneumonia (coronavirus or bacterial infection) admitted to the Intensive Care Unit: Study patients with pneumonia and requirement for oxygen supplementation to achieve oxygen saturation greater than 92% were followed-up, and temperature sensors were be used to register temperature changes in expired air. Clinical evolution of these patients was recorded.
  Interventions: Device: Temperature sensors located in the Venturi mask, placed around the nose and mouth

INTERVENTIONS:
Device: Temperature sensors located in the Venturi mask, placed around the nose and mouth — Temperature sensors from the SC50 series were used, with a single use for each patient. The signals from these sensors were recorded in the supine position with the head elevated at 30º, if possible while the patient was at rest and silent. Simultaneous recordings were be made using the BIOPAC MP 160 system with general-purpose amplifiers (DA 100C).

SUMMARY:
Surveillance and monitoring of patients with respiratory failure before or after undergoing mechanical ventilation is an underdeveloped area compared to the many possibilities of monitoring other non-invasive vital signs that we currently have.

Severe respiratory failure usually affects oxygenation and ventilation. Continuous or frequent non-invasive monitoring of oxygenation is performed with pulse oximetry, with a margin of error between 1 and 4% of arterial oxygen saturation of hemoglobin. Ventilation cannot be fully monitored in non-intubated patients: Measurement of respiratory rate (RR) outside the Intensive Care Unit (ICU) is usually performed intermittently and manually by the nurse, often with a wide margin of error and, regarding tidal volume (VT), it cannot currently be monitored either directly or indirectly in non-intubated patients because the measurement itself interferes with respiration. Similarly, data on inspiratory and expiratory flows cannot be obtained, which are also altered in certain pathologies. The technique considered as a "gold standard" is spirometry, which requires the collaboration of the patient, and the interpretation of the results depends on the performance of the technique in a standardized way. Spirometry offers a single value; continuous monitoring is not feasible and due to the bias of the technique.

More studies are needed to rule out the existence of different breathing patterns of acute respiratory failure and to identify outcome differences between them before recommending different support or treatment approaches.

In a preliminary not published study conducted with healthy volunteers, a good correlation was observed between changes in temperature inside the Venturi mask using two TSC50 thermistors and breathing pattern recorded by thoracic and abdominal plethysmographic bands.

HYPOTHESES: Monitoring respiratory activity, including both RR and the respiratory pattern (tidal volume, inspiratory flow, and the inspiration-to-expiration ratio), could enable early detection of respiratory patterns associated with the worsening of patients with COVID-19 pneumonia and severe pneumonia of other origins.

OBJECTIVES

Main Objective:

To evaluate the ability of the respiratory pattern to early detect respiratory deterioration in patients hospitalized pneumonia before requiring mechanical ventilation.

Specific Objectives:

To describe the initial respiratory pattern and its evolution throughout the hospital stay of patients with acute respiratory failure caused by SARS-CoV-2.

To describe the evolution of the respiratory pattern in patients with bacterial pneumonia admitted to the hospital who require supplemental oxygen.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of COVID-19 pneumonia, community-acquired or hospital-acquired with moderate, severe, or critical severity criteria as defined by the World Health Organization, OR Diagnosis of presumably bacterial pneumonia FINE III, IV or V
* Requirement for oxygen supplementation to achieve oxygen saturation (SpO2) greater than 92%
* Signed informed consent.

Exclusion Criteria:

* Non-invasive ventilation or mechanical ventilation at the time of evaluation
* Chronic noninvasive ventilation or oxygen therapy
* Inclusion in experimental treatment studies where the administered treatment is unknown
* Other more plausible cause of acute respiratory failure (ARF)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with pneumonia admitted to the Intensive Care Unit, requiring oxygen supplementation to achieve an oxygen saturation (SpO2) greater than 92%.
Sampling Method: Non-Probability Sample
Enrollment: 82 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Clinical evolution outcome | From admission to the Intensive Care Unit until discharge or unfavorable outcome, whichever come first , assessed up to two weeks.
  An unfavorable outcome was defined whenever the patient presented with any of the following:
  * PaO2/FiO2 less than 100
  * initiation of High-flow Nasal Oxygen Therapy, or invasive or noninvasive mechanical ventilation
  * death Otherwise the outcome was considered as favorable.

CONTACTS AND LOCATIONS:
Locations (1):
- Complex Hospitalari Universitari Moisès Broggi, Consorci Sanitari Integral, Sant Joan Despí, Barcelona, Spain